CLINICAL TRIAL: NCT01760057
Title: Randomized Controlled Trial to Evaluate the Effect of a Novel Web-based Intervention to Increase HIV Testing in Men Who Have Sex With Men in Lima-Peru
Brief Title: Evaluating the Effect of a Novel Web-based Intervention to Increase HIV Testing in Men Who Have Sex With Men
Acronym: TuNexo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); NGO Via Libre (Other)
Responsible Party: Principal Investigator, Magaly Blas, Research professor, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R01TW008398 (NIH)
Record Dates: First submitted 2012-12-28; First posted 2013-01-03 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: HIV Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health promotion message (Placebo Comparator): Standard online message with an invitation for free HIV testing similar in content to other Peruvian websites
  Interventions: Behavioral: Standard online message with an invitation for free HIV testing similar in content to other Peruvian websites
- Combined Web-based HIV intervention (Experimental): Online HIV testing motivational videos and messages sent via mobile-phone text messaging, e-mail or instant messaging
  Interventions: Behavioral: Online HIV testing motivational videos and messages sent via mobile-phone text messaging, e-mail or instant messaging

INTERVENTIONS:
Behavioral: Online HIV testing motivational videos and messages sent via mobile-phone text messaging, e-mail or instant messaging
  Arms: Combined Web-based HIV intervention
Behavioral: Standard online message with an invitation for free HIV testing similar in content to other Peruvian websites
  Arms: Health promotion message

SUMMARY:
The proposed study is designed to develop and test the effectiveness of a novel web-based HIV intervention to motivate HIV testing among men who have sex with men (MSM). The intervention arm includes the delivery of videos tailored to the reasons MSM have for not getting tested for HIV, as well as HIV testing motivational messages sent via mobile-phone text messaging, e-mail or instant messaging. The intervention and assessments will be guided by the Information-Motivation-Behavioral skills model, the Health Belief Model and the Stages of Change theory. The control intervention will be a health promotion message (similar in content to other Peruvian websites) with an invitation for free HIV testing. Testing will be offered at the Via Libre and Epicentro clinic, and at a mobile unit whose location will be determined based on participants' demand. The outcomes evaluated will be intention to get tested and actual HIV testing among MSM of each of the trial arms.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years of age or older,
* be a man and report having had sex with a man within the last 12 months,
* be a resident of metropolitan Lima, Peru,
* have not been tested for HIV within the last 12 months,
* have a valid e-mail address,
* do not report being HIV positive.

Exclusion Criteria:

* Do not meet the inclusion criteria specified above

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
HIV testing | 6 months after been exposed to the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Magaly M Blas, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (1):
- Universidad Peruana Cayetano Heredia, Lima, Lima Province, Peru

REFERENCES:
- [Background] Blas MM, Alva IE, Cabello R, Carcamo C, Kurth AE. Risk behaviors and reasons for not getting tested for HIV among men who have sex with men: an online survey in Peru. PLoS One. 2011;6(11):e27334. doi: 10.1371/journal.pone.0027334. Epub 2011 Nov 9. PMID 22096551
- [Background] Blas MM, Alva IE, Carcamo CP, Cabello R, Goodreau SM, Kimball AM, Kurth AE. Effect of an online video-based intervention to increase HIV testing in men who have sex with men in Peru. PLoS One. 2010 May 3;5(5):e10448. doi: 10.1371/journal.pone.0010448. PMID 20454667
- [Background] Blas MM, Alva IE, Cabello R, Garcia PJ, Carcamo C, Redmon M, Kimball AM, Ryan R, Kurth AE. Internet as a tool to access high-risk men who have sex with men from a resource-constrained setting: a study from Peru. Sex Transm Infect. 2007 Dec;83(7):567-70. doi: 10.1136/sti.2007.027276. Epub 2007 Oct 11. PMID 17932128
- [Background] Curioso WH, Blas MM, Nodell B, Alva IE, Kurth AE. Opportunities for providing web-based interventions to prevent sexually transmitted infections in Peru. PLoS Med. 2007 Feb;4(2):e11. doi: 10.1371/journal.pmed.0040011. PMID 17326701
- [Result] Blas MM, Menacho LA, Alva IE, Cabello R, Orellana ER. Motivating men who have sex with men to get tested for HIV through the internet and mobile phones: a qualitative study. PLoS One. 2013;8(1):e54012. doi: 10.1371/journal.pone.0054012. Epub 2013 Jan 8. PMID 23320116